CLINICAL TRIAL: NCT06331884
Title: Phase 1 Study on the Safety, Tolerability and Pharmacokinetics/-Dynamics of Escalating Single Intravenous Doses of AK1967 (Procizumab) in Healthy Male Volunteers
Brief Title: Phase 1 Study to Evaluate Safety, Tolerability and Pharmacokinetics/-Dynamics of AK1967 (Procizumab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4TEEN4 Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCZ_Phase1
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Safety and Tolerability; Healthy Volunteers
MeSH Terms: interventions — procizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AK1967 3 mg/kg/body weight (Active Comparator)
  Interventions: Drug: AK1967 (Procizumab)
- AK1967 6 mg/kg/body weight (Active Comparator)
  Interventions: Drug: AK1967 (Procizumab)
- AK1967 12 mg/kg/body weight (Active Comparator)
  Interventions: Drug: AK1967 (Procizumab)

INTERVENTIONS:
Drug: AK1967 (Procizumab) — DPP3 inhibition using the humanized monoclonal antibody AK1967 (Procizumab)
  Arms: AK1967 12 mg/kg/body weight; AK1967 3 mg/kg/body weight; AK1967 6 mg/kg/body weight
Drug: Placebo — Application of placebo
  Arms: Placebo

SUMMARY:
Dipeptidyl peptidase 3 (DPP3) is a protease involved in the degradation of several cardiovascular mediators. During cardiogenic shock, upregulation of the vasoconstrictive molecule angiotensin II is a physiologic and potentially life-saving response aimed at maintaining adequate tissue perfusion. As circulating (c)DPP3 is able to effectively cleave angiotensin II, it may represent a novel factor contributing to hemodynamic instability during cardiogenic shock.

Recently, a cDPP3-antagonizing antibody called AK1967 (commonly referred to as Procizumab) has been developed. In animal models of cardiogenic- and septic shock, inhibition of cDPP3 by AK1967 resulted in improved cardiac function and survival. Furthermore, AK1967 has shown an excellent safety record in different preclinical studies. In the current study the safety, tolerability and pharmacokinetics/-dynamics of AK1967 will be investigated in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this trial prior to any study-mandated procedure.
* Male subjects aged 18 to 35 years inclusive.
* Subjects have to agree to use a reliable way of contraception with their partners from study entry until one month after study drug administration.
* BMI between 18 and 30 kg/m², with a lower limit of body weight of 50 kg and an upper limit of 100 kg.
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram, and clinical laboratory parameters.

Exclusion Criteria:

* Unwillingness to abstain from any medication, including recreational drugs or vitamin supplements during the course of the study and within two days prior to the treatment day.
* Unwillingness to abstain from alcohol within one day prior to the treatment day until one day after the treatment day.
* Surgery or trauma with significant blood loss or blood donation within one month prior to the treatment day.
* History, signs or symptoms of cardiovascular disease, in particular:

  * History of frequent vasovagal collapse or of orthostatic hypotension
  * Resting pulse rate ≤45 or ≥100 beats/min
  * Hypertension (RR systolic >160 or RR diastolic >90 mmHg)
  * Hypotension (RR systolic <100 or RR diastolic <50 mmHg)
  * Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
  * Any chronic cardiac arrhythmias (except PAC's, PVC's)
* Renal impairment: plasma creatinine >120 μmol/L
* Liver function tests (alkaline phosphatase, AST, ALT and/or γ-GT) above 2x the upper limit of normal.
* History of asthma
* Atopic constitution
* CRP above 2x the upper limit of normal, or clinically significant acute illness, including infections, within two weeks prior to the treatment day.
* Treatment with investigational drugs or participation in any other clinical trial within 30 days prior to the treatment day.
* Known or suspected of not being able to comply with the trial protocol.
* Known hypersensitivity or allergic reactions to drug compounds, (i.e. previous adverse drug reactions).
* Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single intravenous infusion of placebo (vehicle solution matching AK1967) over a 2-hour period
- AK1967 3 mg/kg/Body Weight: Single intravenous infusion of AK1967 (Procizumab) at a dose of 3 mg/kg over a 2-hour period
- AK1967 6 mg/kg/Body Weight: Single intravenous infusion of AK1967 (Procizumab) at a dose of 6 mg/kg over a 2-hour period
- AK1967 12 mg/kg/Body Weight: Single intravenous infusion of AK1967 (Procizumab) at a dose of 12 mg/kg over a 2-hour period
Period: Overall Study
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Number of adverse events (AEs)
Time Frame: 28 days
Measure: Number; unit: AEs
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight
Number analyzed (Participants) | 6 | 6 | 6 | 6
AEs | 7 | 8 | 12 | 3

2. Secondary Outcome: Pharmacokinetics of AK1967 - t1/2
Description: Pharmacokinetics of AK1967 - t1/2 (Half life)
Time Frame: 28-days
Population: PK measurements were done in all arms, however for the participants from the placebo group, the measurement results was below the "Lower Limit of Quantification".
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight
Number analyzed (Participants) | 6 | 6 | 6 | 6
h | NA (NA) — Measurement results was below Lower Limit of Quantification | 24.3 (2.81) | 34.3 (16.6) | 53.1 (21.5)

3. Secondary Outcome: Pharmacokinetics of AK1967 - AUC
Description: Pharmacokinetics of AK1967 - Area Under the Curve
Time Frame: 28 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µg*h/ml
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight
Number analyzed (Participants) | 6 | 6 | 6 | 6
µg*h/ml | NA (NA) — Measurement results was below Lower Limit of Quantification | 345 (67.9) | 845 (336) | 2076 (584)

ADVERSE EVENTS:
Time Frame: From start of IMP administration up until the last follow up visit 28 days after IMP administration
Arm/Group | Placebo | AK1967 3 mg/kg/Body Weight | AK1967 6 mg/kg/Body Weight | AK1967 12 mg/kg/Body Weight
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | AK1967 3 mg/kg/Body Weight (N=6) | AK1967 6 mg/kg/Body Weight (N=6) | AK1967 12 mg/kg/Body Weight (N=6)
Sore throat and nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Headache and neckpain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
headache, combined with symptoms of exhaustion (General disorders) | 1 | 0 | 0 | 0
Episodic stinging pain around the left collarbone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tonsilitis accompanied by a fever and fatigue (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
shooting pains in the left flank (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Slight burning sensation in right arm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Itchy nose, itchy and red eyes (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Soreness and a hematoma on the place of a failed arterial catheterization (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Normocytemic anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Nasal congestion and irritated eyes (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Feeling of some pressure in outlet of catheters (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sore throat, runny nose and swollen glands (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Swollen and painfull left knee (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Runny nose and itchy eyes (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Increased frequency of bruising (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Light headed feeling with getting up (Nervous system disorders) | 0 | 0 | 1 | 0
Knee pain (left) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Nose bleeds (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Shortness of breath, which subject attributes to (known) asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tiredness, headache (General disorders) | 1 | 0 | 0 | 0
Accident (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Diarrhea and vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Infection finger (Infections and infestations) | 0 | 0 | 0 | 1
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT06331884/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT06331884/SAP_001.pdf